CLINICAL TRIAL: NCT04085172
Title: A Phase 4, Multicenter, 2-part Study Composed of a Randomized, Double-blind, Parallel-group, Placebo-controlled, Active-comparator, Dose-optimization Evaluation Followed by a 1-Year Open-label Evaluation to Assess the Safety and Efficacy of Guanfacine Hydrochloride Prolonged-release (SPD503) in Children and Adolescents Aged 6 to 17 Years With Attention-deficit/Hyperactivity Disorder
Brief Title: A Study of TAK-503 in Children and Teenagers With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD503-401; 2018-000821-29 (EudraCT Number); TAK-503-401 (Other: Takeda Development Center Americas, Inc.); 2022-502630-71-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study contains two parts (Part A and Part B), where Part A will be double blind, double dummy parts of the study followed by Part B as an open label part of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Guanfacine hydrochloride (TAK-503) (Experimental): Participants randomized to TAK-503 will receive initial dose of 1 milligram (mg), and up titrated with weekly incremental dose of 1 mg until an optimal dose is reached. Participants aged 6 to 12 years will receive a dose of 1 to 4 mg and aged 13 to 17 years will receive a dose of 5 to 7 mg TAK-503 oral tablet once daily (QD) for 18 weeks.
  Interventions: Drug: Guanfacine hydrochloride (TAK-503)
- Part A: Atomoxetine hydrochloride (Active Comparator): Participants who weigh less than (<) 70 kilograms (kg) at baseline will receive Atomoxetine hydrochloride capsule orally at an initial dose of 0.5 milligram per kilogram (mg/kg) which may be increased to the target dose of 1.2 mg/kg oral capsule QD during the treatment of 18 weeks. Permitted doses of Atomoxetine hydrochloride capsule will be 10, 18, 25, 40, 60, and 80 mg QD. Participants who weigh >= 70 kg at baseline will receive Atomoxetine hydrochloride at an initial dose of 40 mg oral capsule QD which may be increased to 80 mg and then to 100 mg for 18 weeks. The total dose for participants who weigh >= 70 kg at baseline will not exceed 100 mg.
  Interventions: Drug: Atomoxetine hydrochloride
- Part A: Placebo (Placebo Comparator): Participants aged 6 to 12 years will receive a dose of 1 to 4 mg tablet of placebo matched to TAK-503 and aged 13 to 17 years will receive a dose of 5 to 7 mg tablets of placebo matched to TAK-503 orally QD for 18 weeks. Participants who weigh < 70 kg at baseline will receive placebo matched to Atomoxetine hydrochloride oral capsule at an initial dose of 0.5 mg/kg which may be increased to the target dose of 1.2 mg/kg QD oral capsule during the treatment of 18 weeks. Permitted doses of placebo matched to Atomoxetine hydrochloride will be 10, 18, 25, 40, 60, and 80 mg QD and participants who weigh >= 70 kg will receive placebo matched to Atomoxetine hydrochloride at an initial dose of 40 mg QD capsule orally which may be increased to 80 mg and then to 100 mg.
  Interventions: Other: Placebo
- Part B: Guanfacine hydrochloride (TAK-503) (Experimental): Participants from Part A will roll over into Part B directly after 18 weeks and will receive TAK-503 at an initial dose of 1 mg, and up titrated with weekly incremental dose of 1 mg until an optimal dose is reached. Participants aged 6 to 12 years will receive a dose of 1 to 4 mg and aged 13 to 17 years will receive a dose of 5 to 7 mg TAK-503 oral tablet QD for 52 weeks of Part B.
  Interventions: Drug: Guanfacine hydrochloride (TAK-503)

INTERVENTIONS:
Drug: Guanfacine hydrochloride (TAK-503) — Participants aged 6 to 12 years will receive a dose of 1 to 4 mg and aged 13 to 17 years will receive a dose of 5 to 7 mg TAK-503 oral tablets once daily for 18 weeks in Part A or 52 weeks in Part B.
  Other Names: Intuniv; SPD503
  Arms: Part A: Guanfacine hydrochloride (TAK-503); Part B: Guanfacine hydrochloride (TAK-503)
Drug: Atomoxetine hydrochloride — Participants will receive Atomoxetine hydrochloride oral capsule once daily for 18 weeks in Part A.
  Arms: Part A: Atomoxetine hydrochloride
Other: Placebo — Participants aged 6 to 12 years will receive a dose of 1 to 4 mg and aged 13 to 17 years will receive a dose of 5 to 7 mg placebo matched to TAK 503 oral tablets once daily for 18 weeks and placebo matched to atomoxetine hydrochloride oral capsules at once daily for 18 weeks in Part A.
  Arms: Part A: Placebo

SUMMARY:
The main aim of this study is learn more about long-term TAK-503 treatment in children and teenagers with ADHD for whom earlier stimulant treatment did not work.

The study has two parts (A and B). In Part A, participants will take tablets of TAK-503, atomoxetine or placebo and in Part B TAK-503 tablets.

DETAILED DESCRIPTION:
This study will be conducted in two parts Part A and Part B. Part A is a double-blinded, double-dummy, placebo-controlled study with an atomoxetine arm as an active reference to TAK-503. Eligible participants with ADHD will be randomized in a 1:1:1 ratio among TAK-503, atomoxetine, and placebo treatment arms for 18 weeks of double-blinded treatment. At the end of the 18 weeks, participants will roll over to Part B directly as per the study protocol directions for an additional 52 weeks of open-label TAK-503 treatment.

ELIGIBILITY:
Inclusion Criteria:

Study Part A:

* Participant is a male or female aged 6 to 17 years inclusive at the time of consent/assent.
* Participant must meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation using the Kiddie-Schedule for Affective Disorders-Present and Lifetime Version (K-SADS-PL) by a trained child and adolescent psychiatrist at screening (Visit 1A).
* Participant for whom prior stimulant therapy is not suitable, not tolerated, or shown to be ineffective as determined by investigator clinical assessment and review of the Prior Stimulant Medication Questionnaire (PSMQ) administered during screening (Visit 1A).
* Participant has an ADHD-RS-5 total score greater than or equal to (> =) 28 at baseline (Visit 2A).
* Participant has a baseline (Visit 2A) CGI-S score > = 4.
* Participant who is a female of childbearing potential (FOCP) and postmenarchal must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at screening (Visit 1A) and a negative urine pregnancy test at baseline (Visit 2A), be nonlactating, and agree to comply with any applicable contraceptive requirements described in the protocol. Female of child bearing potential is defined as any female participant who is at least aged 9 years or younger than 9 years and postmenarchal.
* Participants parent or legally authorized representative (LAR) must provide signature of informed consent. Documentation of assent (if applicable) must be provided by the participant indicating that the participant is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6[R2] and applicable regulations, before completing any study-related procedures.
* Participant and parent/LAR are willing and able to comply with all the testing and requirements defined in this protocol, including oversight of morning dosing. Specifically, the parent/LAR must be available for the duration of the study to administer the investigational medicinal product (IMP) dose each morning when the participant awakens.
* Participant has supine and standing blood pressure (BP) measurements less than the 95th percentile for age, sex, and height at both screening (Visit 1A) and baseline (Visit 2A).
* Participant is functioning at an age-appropriate level intellectually, as judged by the investigator.
* Participant is able to swallow intact tablets and capsules.

Study Part B:

* Female participants of child-bearing potential must have a negative serum β-hCG pregnancy test if a screening visit is conducted and/or a negative urine pregnancy test at baseline and agree to comply with any applicable contraceptive requirements of the protocol. An FOCP is defined as any female participant who is at least aged 9 years or younger than 9 years and postmenarchal.
* Participant has a supine and standing BP measurement less than the 95th percentile for age, sex, and height.

Exclusion Criteria:

Study Part A:

* Participant has a current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder (except oppositional defiant disorder), including but not limited to any of the following comorbid Axis I and Axis II disorders (the K-SADS-PL should be reviewed to confirm diagnosis, if necessary):

  1. Post-traumatic stress disorder (PTSD)
  2. Bipolar illness, psychosis, or family history in either biological parent
  3. Pervasive developmental disorder
  4. Obsessive-compulsive disorder (OCD)
  5. Psychosis/schizophrenia
  6. Serious tic disorder or a family history of Tourette's disorder
* Participant is currently considered to be a suicide risk by the investigator; has made a previous suicide attempt; has a history of, or currently demonstrating, active suicidal ideation.
* Participant has a substance abuse disorder as defined by DSM-5 criteria or has been suspected of a substance abuse or dependence disorder (except nicotine) within the past 6 months.
* Participant has a clinically important abnormality on the urine drug and alcohol screen (except for the participants current ADHD stimulant, if applicable) at screening (Visit 1A).
* Participant has been physically, sexually, and/or emotionally abused.
* Participant has any other disorder that as judged by the investigator could contraindicate TAK-503 or confound the results of the safety and efficacy assessments.
* Participant has any condition or illness including any clinically significant abnormal laboratory value at screening (Visit 1A) or, if the laboratory test was repeated, at baseline (Visit 2A) that, as judged by the investigator, would be an inappropriate risk to the participant and/or could confound the interpretation of study results.
* Participant has current abnormal thyroid function, defined as abnormal thyroid-stimulating hormone and thyroxine at screening (Visit 1A). Treatment with a stable dose of thyroid medication for > = 3 months before screening will be permitted.
* Participant has a known history or presence of: malignancy (except nonmelanoma skin cancer), pregnancy, and/or a developmental delay or abnormality associated with growth or sexual maturation delays that are not related to ADHD.
* Children aged 6 to 12 years with a body weight less than (<) 25.0 kg or adolescents aged > = 13 years with a body weight < 34.0 kg at screening (Visit 1A) or baseline (Visit 2A).
* Participant is significantly overweight based on the Centers for Disease Control (CDC) BMI-for-age sex-specific charts at screening (Visit 1A) or baseline (Visit 2A). For this study, significantly overweight will be defined as a BMI that is greater than the 95th percentile.
* Participant has a known history or presence of: structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (e.g. clinically significant heart block or QT interval prolongation), bradycardia, or exercise-related cardiac events including syncope and presyncope.
* Participant has clinically significant electrocardiogram (ECG) findings, as judged by the investigator, at baseline (Visit 2A).
* Participant has orthostatic hypotension* or a known history of hypertension. (*Orthostatic hypotension is defined as a sustained reduction of systolic blood pressure of at least 20 millimeter of mercury (mm Hg) or diastolic blood pressure of 10 mm Hg within 3 minutes of standing from supine.)
* Participant has a known family history of sudden cardiac death or ventricular arrhythmia.
* Participant is currently using any medication that violates protocol-specified washout criteria at baseline (Visit 2A), including any ADHD medication or other prohibited medications such as herbal supplements, medications that affect BP or heart rate (HR) or medications that have central nervous system (CNS) effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications (i.e., antihistamines).
* Participant has a medical condition except ADHD that requires treatment with any medication that affects the CNS.
* Participant is female and pregnant or currently lactating.
* Participant has taken another investigational product or participated in a clinical study within 30 days before screening (Visit 1A).
* Participant does not tolerate or has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride, atomoxetine, or any TAK-503 or atomoxetine drug product component.
* Participant has a history of a seizure disorder (except for a single childhood febrile seizure episode that occurred before the age of 3 years)
* Participant is well-controlled on his/her current ADHD medication with acceptable tolerability, and the parent/treating physician does not object to the current medication.
* Participant has alanine transaminase (ALT) greater than (>) 2*upper limit of normal (ULN) or aspartate aminotransferase (AST) >2*ULN or bilirubin >1.5*ULN at screening.

Study Part B:

* Participant failed screening, voluntarily withdrew, or was discontinued from Study Part A for protocol nonadherence, participant noncompliance, or TEAE or SAE.
* Participant had any clinically significant TEAE during Study Part A that, as judged by the investigator, would preclude exposure to TAK-503.
* Participant has a history of alcohol or other substance abuse or dependence, as defined by DSM-5 (with the exception of nicotine) within the last 6 months.
* Participant currently uses any of the prohibited medication or other medications, including herbal supplements, that affect BP or HR or that have CNS effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications (i.e. antihistamines) in violation of the protocol-specified washout criteria at baseline.
* Participant has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride, or any components found in TAK-503.
* Participant has taken any IMP except placebo in Study Part A within the 30 days before baseline of Study Part B (Visit 2B).
* Participant is significantly overweight based on the CDC BMI-for-age sex-specific charts at screening. Significantly overweight is defined as a BMI > 95th percentile.
* Participant is a child aged 6 to 12 years with a body weight of < 25.0 kg or an adolescent aged > = 13 years with a body weight of < 34.0 kg at screening (Visit 1B)
* Participant has any condition or illness including clinically significant abnormal laboratory values at screening which as judged by the investigator would represent an inappropriate risk to the participant and/or confound the interpretation of study results.
* Participant is currently considered a suicide risk as judged by the investigator, has previously made a suicide attempt, has a history of, or is currently demonstrating active suicidal ideation. Participants with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the investigator.
* Participant has clinically significant ECG findings, as judged by the investigator, at baseline (Visit 2B).
* Participant has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (e.g. clinically significant heart block), exercise-related cardiac events including syncope and presyncope, or clinically significant bradycardia.
* Participant has orthostatic hypotension or a known history of hypertension. (*Orthostatic hypotension is defined as a sustained reduction of systolic blood pressure of at least 20 mm Hg or diastolic blood pressure of 10 mm Hg within 3 minutes of standing from supine).
* Participant has a history of a seizure disorder (except for a single childhood febrile seizure episode that occurred before the age of 3 years) or the presence of a serious tic disorder including Tourette's syndrome.
* Participant has a medical condition except ADHD, which requires treatment with any medication that affects the CNS.
* Participant has ALT >2*ULN or AST >2*ULN or bilirubin >1.5*ULN at screening.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Change From Baseline in the Reaction Time (RTI) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Week 10 | Baseline, Week 10
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. The RTI task of CANTAB involves elements of decision-making and attention as measured by choice accuracy as well as motor responses, by measuring motor and mental response speeds, and assesses movement time, reaction time, response accuracy, and impulsivity. This outcome measure will be assessed at Week 10 in both Part A and Part B of the study.
Part A: Change from Baseline in the Reaction Time (RTI) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Week 18 | Baseline, Week 18
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. The RTI task of CANTAB involves elements of decision-making and attention as measured by choice accuracy as well as motor responses, by measuring motor and mental response speeds, and assesses movement time, reaction time, response accuracy, and impulsivity. This outcome measure will be assessed at Week 18 in Part A of the study.
Part B: Change From Baseline in the Reaction Time (RTI) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Week 49 | Baseline, Week 49
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. The RTI task of CANTAB involves elements of decision-making and attention as measured by choice accuracy as well as motor responses, by measuring motor and mental response speeds, and assesses movement time, reaction time, response accuracy, and impulsivity. This outcome measure will be assessed at Week 49 in Part B of the study.

SECONDARY OUTCOMES:
Parts A and B: Change From Baseline in the Rapid Visual Information Processing (RVP) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Specified Time Points | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 49
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. Cognitive domain, sustained attention will be measured by the CANTAB RVP task. RVP measures the ability to sustain attention over time and is a sensitive measure of frontal-parietal function. In this task, single digits appear in a pseudo-random order at a rate of 100 digits per minute in a box at the center of the screen. Participants are to detect a 3-digit target sequence (e.g. 2-4-6) and respond by pressing a button at the bottom of the screen when the final number of the sequence appears on the screen.
Parts A and B: Change From Baseline in the Spatial Working Memory (SWM) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Specified Time Points | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 49
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments, SWM is a component of cognitive executive function which is measured by SWM task of CANTAB between the errors. The ability to retain spatial information and manipulate remembered items in working memory will be measured with the SWM task of CANTAB which is self-ordered and assesses the individual's ability to strategize heuristically. The test is a sensitive measure of frontal lobe and executive dysfunction.
Parts A and B: Change From Baseline in the Stop Signal Task (SST) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Specified Time Points | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 49
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. Response control or inhibition cognitive domain will be measured by the CANTAB SST. SST measure response inhibition. The participant must respond to an arrow stimulus by touching either of 2 choices depending on the direction the arrow points. If an audio tone is present, the participant is not to respond.
Parts A and B: Change From Baseline in the Delayed Matching to Sample (DMS) Task of the Cambridge Automated Neuropsychological Test Battery (CANTAB) at Specified Time Points | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 49
  The neurocognitive function effects of TAK-503 on adolescents and children diagnosed with ADHD will be evaluated using the CANTAB cognitive assessments. Recognition memory of cognition domain will be measured by the CANTAB DMS task. DMS measures both simultaneous matching and short-term visual memory. The participant is shown a complex visual pattern (the sample) and after a brief delay, 4 similar patterns. The participant must identify the pattern that matches the sample.
Parts A and B: Tanner Stage at Specified Time Points | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 49
  Sexual maturation will be measured by Tanner stage. The stage of puberty or sexual maturation will be evaluated for each participant according to Tanner staging. The Tanner stage for genitals (male, stages I-V), breasts (females, stages I-V), and pubic hair (both sexes, stages I-V) will be documented at the specified times. Tanner staging will be self-assessed. Self-assessment in this study is defined as participants or parents indicating which drawing of the scale corresponds to participants sexual maturation stage at the time of the specific visit.
Parts A and B: Number of Participants With Clinically Significant Changes in Vital signs, ECG, Physical Examination | Part A: From start of study drug administration up to Week 18; Part B: From start of study drug administration up to follow up (Week 53)
  Physical examinations will include height and weight. Growth will be measured by weight, height, and BMI. Body mass index is a measure of body fat based on height and weight. Vital signs will be assessed based on blood pressure, pulse rate, respiratory rate and body temperature in both Part A and Part B. The HR, PR interval, QRS interval, and QT interval will be measured from all ECGs and the QTcB and QTcF assessed at specified time points in both Part A and Part B of the study.
Parts A and B: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Part A: From start of study drug administration up to Week 18; Part B: From start of study drug administration up to follow up (Week 53)
  An Adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with an investigational product or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the investigational product or medicinal product. TEAEs include both serious and non-serious AEs.
Parts A and B: Brief Psychiatric Rating Scale for Children (BPRS-C) | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36 and Week 49
  Psychiatric symptoms will be measured by the Brief Psychiatric Rating Scale for Children (BPRS-C) total score. The 21 items of the clinician-rated BPRS-C are grouped into the following 7 scales: depression, anxiety, psychomotor excitation, behavior problems, withdrawal, thinking disturbance, and organicity. Each item of the 21 items is clinician-graded using the following 7-point severity Likert-scale from 0 to 6 (not present=0; very mild=1; mild=2; moderate=3; moderately severe=4; severe=5; extremely severe=6. BPRS-C will be assessed at specified time points in both Part A and Part B.
Parts A and B: Columbia- Suicide Severity Rating Scale (CSSRS) | Part A: Baseline (from start of study drug administration) up to Week 18; Part B: Baseline (from start of study drug administration) to Week 52
  The C-SSRS is a structured tool to assess suicidal ideation and behavior. A maximum of 19 items will be completed as follows: 7 items are required, a potential 10 additional items will be completed upon a positive response to a required item, and 2 items completed if suicide or suicide-like behavior is observed during the interview. The C-SSRS uses dichotomous scales (i e, yes or no), Likert scales, and text or narrative to further describe thoughts or behaviors. C-SSRS Score will be assessed at specified time points in both Part A and Part B.
Parts A and B: Udvalg for Kliniske Undersøgelser (UKU) Side Effect Rating Scale | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36, Week 49, Week 50, Week 51 and Week 52
  UKU rating scale was developed for clinicians to assess side effects of psychopharmacological medications based on interviews and other relevant source information. UKU items relevant to the established safety profile of TAK-503 such as Increased Duration of Sleep, Asthenia or Lassitude or lncreased Fatigability, Sleepiness or Sedation, and Orthostatic Dizziness. UKU rating scale will be assessed at specified time points in both Part A and Part B.
Parts A and B: Pediatric Daytime Sleepiness Scale (PDSS) | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36 and Week 49
  Sedative effects will be measured by participant ratings on the Pediatric Daytime Sleepiness Scale (PDSS). The PDSS is a self-reported assessment of daytime sleepiness in children aged 11 to 15 years. PDSS questionnaire was designed to be easy to administer, score, and interpret. Sleepiness-related questions are based on previous research of situations that can be sensitive to sleep loss in this age group. The 8 questions are scored on Likert-scale from 0 to 4 (never=0; seldom=1; sometimes=2; frequently=3; always=4). The total score on the PDSS can range from 0 (never sleepy) to 32 (always sleepy). PDSS will be assessed at specified time points in both Part A and Part B.
Parts A and B: ADHD-Rating Scale-5 (ADHD-RS-5) Total Score and Subscales | Part A: Baseline, Week 1, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36 and Week 49
  The ADHD-RS-5 (DuPaul et al., 2016) is used widely by mental health, educational, and medical practitioners in screening, diagnosis, and treatment evaluation to determine the frequency and severity of ADHD symptoms and impairments in children and adolescents. Attention-deficit/hyperactivity disorder symptoms is measured by the investigator-administered ADHD-Rating Scale-5 (ADHD-RS-5) total score and hyperactivity/impulsivity and inattention symptoms as subscale scores. The ADHD-RS-5 is based on the diagnostic criteria for ADHD as described in the DSM-5 and consists of 2 symptom subscales, inattention and hyperactivity-impulsivity, each with 9 items and a total scale of 18 items. Each item in the subscale is scored with a value ranging from 0 (no symptoms) to 3 (severe symptoms). The total score can range from 0 to 54. ADHD-RS-5 Total Score and Subscales wiil be assessed at specified time points in both Part A and Part B.
Parts A and B: Clinical Global Impression-Improvement (CGI-I) | Part A: Week 1, Week 10, Week 18 Part B: Week 10, Week 23, Week 36 and Week 49
  Global clinical measurement of ADHD improvement as measured by Clinical Global Impression-Improvement (CGI-I) using the Clinical Global Impression-Severity (CGI-S) to establish baseline. The CGI scale will be used to evaluate the severity of mental illness over time. The CGI-S will be administered to assess the severity of mental illness at baseline. The CGI-S is scored on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The CGI-I is also scored on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). CGI-I will be measured at specified time points in both Part A and Part B.
Parts A and B: Child Health and Illness Profile - Child Edition: Parent Report Form (CHIP-CE:PRF) | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36 and Week 49
  The Parent Report Form of the Child Health and Illness Profile - Child Edition (CHIP-CE:PRF) will be administered to provide information on self-esteem and school functioning in pediatric participants diagnosed with ADHD. The 5 domains and 12 subdomains covered in the 76 items comprising the CHIP-CE:PRF. Satisfaction: with health (7 items) and self (4 items); Comfort: physical (9 items) and emotional symptoms (9 items) and activity restrictions (4 items) due to illness; Resilience: behaviors and family involvement (8 items) in activities likely to enhance health, Social problem-solving (5 items),Physical activity (6 items); Risk avoidance: behaviors that if not avoided are likely to pose risks to health: Individual risk avoidance (4 items), Threats to achievement (10 items); Achievement: developmentally appropriate role functioning in school and with peers: Academic performance (5 items), Peer relations (5 items). CHIP-CE: PRF will be assessed in both Part A and Part B.
Parts A and B: Conners 3 Parent Short Form (C3PS) Total Score | Part A: Baseline, Week 10, Week 18 Part B: Baseline, Week 10, Week 23, Week 36 and Week 49
  The Conners 3 is a focused diagnostic tool for the assessment of ADHD and associated learning, behavior, and emotional problems in children 6 to 18 years of age. The C3PS is completed by a child's parent/guardian and is comprised of 45 items with subsets of items related to six content scales: inattention, hyperactivity/impulsivity, executive functioning, learning problems, defiance/aggression and peer relations. The parent rates his/her child on the first 43 items of the C3PS using a 4-point Likert scale (0-3; where 0=not at all true [never, seldom] and 3=very much true [very often, very frequently]) based on past month; the last 2 items are fill-in-the-blank and do not contribute to the raw score(s). Raw scores are converted to T-scores. Lower change from baseline T-scores (<0) represent a better outcome. C3PS Total score will be assessed in both Part A and Part B.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas
Locations (50):
- United States (20):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Advanced Research Center, Inc., Anaheim, California
  - Sun Valley Research Center, Inc., Imperial, California
  - Alliance Research, Long Beach, California
  - PCSD Feighner Research, San Diego, California
  - Homestead Medical Research, Homestead, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Care Research Center, Inc., Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - AMR Conventions Research, Ltd, Naperville, Illinois
  - Collective Medical Research LLC, Prairie Village, Kansas
  - Qualmedica Research, LLC, Bowling Green, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - University of Cincinnati, Cincinnati, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Clinical Research Partners, LLC, Petersburg, Virginia
- Austria (2):
  - LKH-Klinikum Graz, Graz
  - Medizinische Universtität Wien, Vienna
- Belgium (3):
  - UZ Brussel, Brussels
  - UPC KU Leuven Afdeling Kinderpsychiatrie ADHD-raadpleging, Leuven
  - Foyer Saint Francois, Namur
- Germany (4):
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Rheinhessen-Fachklinik Mainz, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Netherlands (2):
  - EB FlevoResearch, Almere Stad
  - EB UtrechtResearch, Utrecht
- Portugal (6):
  - Hospital de Cascais - Dr. José de Almeida, Alcabideche
  - Centro Clinico Academico 2CA Associacao Braga, Hospital de Braga Piso 1, Ala E, Braga
  - Centro Hospitalar Universitario Cova da Beira, E.P.E, Covilha
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - Hospital CUF Descobertas, Lisbon
  - Centro Materno Infantil do Norte (CMIN) Centro Hospitalar Universitario do Porto, Porto
- Spain (8):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Clinica Dr. Quintero, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Complejo Hospitalario de Palencia, Palencia
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Instituto Valenciano de Neurología Pediátrica (INVANEP), Valencia
- Sweden (3):
  - Barnneuropsykiatriska enheten, Sahlgrenska University hospital, Gothenburg
  - Regionhälsan, Mölnlycke
  - PRIMA Barn- och Vuxenpsykiatri AB, Norsborg
- United Kingdom (2):
  - Tayside Children Hospital, Dundee
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b600a4db2bf003ab48b68